CLINICAL TRIAL: NCT05218291
Title: the Effect of Technology Applıed Yoga on Care Load, Qualıty of Lıfe, and Psychologıcal Well-Beıng of Indıvıduals Wıth Specıal Needs
Brief Title: The Effect of Yoga on Care Load, Quality of Life, and Psychological Well-Being of Indivıduals With Special Needs
Acronym: Yoga
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Tuğba Özdemir, research assistant, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 55
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Caregiver Burden; Quality of Life; Psychological Stress
Keywords: yoga; Caregiver burden; Quality of Life; psychological well-being; individuals with special needs
MeSH Terms: conditions — Caregiver Burden; Stress, Psychological; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology-Supported Yoga Applied Group (Experimental): The yoga initiative to be applied to the intervention group; Yoga, which is mind-breath-body work; It includes meditation, pranayama (breath work), and asanas (yoga poses).
  The content of the yoga practice consists of the following poses:
  -Tadasana (Mountain pose), -Urdhvahastasana, -Uttanasana, -Ardha Uttanasana, -Plank, -Ashtang Pranam, -Bhujangasana (Mini cobra), -Adho Mukha Svanasana (Downward facing dog), -Vrksasana (Tree Pose), - Utthita Trikonasana (Triangle Pose), -Virabhadrasana I (Warrior I), -Virabhadrasana II (Warrior II), -Virabhadrasana I with Anjali Mudra (Hands Reverse Namaste), -Utkatasana (Chair Pose), -Salabhasana, -Paschimottanasana , -Dandasana, -Salamba Sarvangasana (Shoulder pose), -Ardha Urdhva Dhanurasana (Half Wheel Pose), -Reverse Warrior, -Child's pose, -Ananda Balasana (Happy baby), -Wipers, -Corpse Pose
  Interventions: Other: Yoga Practice
- Control Group (Active Comparator): No intervention was made in caregivers.
  Interventions: Other: Ongoing caregivers

INTERVENTIONS:
Other: Yoga Practice — In this study, the yoga initiative to be made for the caregivers in the experimental group consists of breathing, meditation and yoga poses.
  Arms: Technology-Supported Yoga Applied Group
Other: Ongoing caregivers — Caregivers included in the control group, who did not apply any yoga intervention, will be observed as caregivers.
  Arms: Control Group

SUMMARY:
The fact that an individual has a physical, social or mental disability affects not only the individual, but also the close environment of the individual and even the society in which he lives. Those who are most affected by this situation in the society are undoubtedly the caregivers. Caregivers of individuals with disabilities experience more anxiety than other caregivers, spare less time for themselves, and participate in less physical and social activities. As a result of social, physical and emotional burdens on parents and other caregivers of disabled individuals, low quality of life, unhealthy family function and negative psychological conditions are observed in caregivers, especially stress. Problems related to financial situation, exclusion from social environment, psychological state, sense of burnout and educational status are among the other problems experienced by caregivers. The aim of this study; The aim of this study is to examine the effects of technology supported yoga applied to caregivers of individuals with special needs on care burden, quality of life and psychological well-being. Research data will be collected from the caregivers of individuals with special needs registered in a Guidance and Research Center in a province. The data of the study will be collected using the Socio-demographic Data Collection Form, the Caregiver Burden Scale, the Multidimensional Quality of Life Scale, and the Warwick-Edinburgh Mental Well-Being Scale. The study is in a randomized controlled design. SPSS 25.0 program will be used in the data analysis of the research. Descriptive data will be analyzed using number, percentage, mean, standard deviations. Spearman test will be applied to determine the correlations between the scale scores. of groups Homogeneity in terms of descriptive statistics will be analyzed with the Kolmogorov Smirnov Test. Student t or Mann Whitney U tests will be used to compare numerical data in two independent groups, and One-way ANOVA or Kruskal Wallis tests will be used for comparisons in more than two independent groups. Relationships between categorical variables will be tested with chi-square test and relationships between numerical variables will be tested with correlation coefficient. The significance level will be accepted as 0.05. The power and effect size of the study will be calculated by regression analysis.

DETAILED DESCRIPTION:
Caregivers mostly consist of parents and even mothers. As primary caregivers in the care of a healthy newborn, mothers experience many physical, emotional and mental problems. Every parent makes plans for their child to be born, their social environment and their own expectations for their children are formed, and therefore, giving birth to a disabled child means that all these planning and expectations are subject to change. Problems related to financial situation, exclusion from social environment, psychological state, sense of burnout and educational status are among the other problems experienced by caregivers. It has been determined that there are many problems that caregivers experience psychologically, and it is necessary to support caregivers by conducting various interventional studies for these problems. As a result of the researches carried out in the caregivers of the disabled individuals, the existence of negative psychological conditions such as low quality of life, depression and anxiety has been determined and it has been seen that interventional studies are needed in this regard. It has been concluded that yoga has positive effects on other caregivers regarding the problems experienced by caregivers of disabled individuals. This study was planned in accordance with the randomized controlled research design. It will be held between November 2021 and April 2022 with the caregivers of the students registered in the Guidance and Research Centers in Gebze and Darıca Districts of Kocaeli Province. All caregivers between the ages of 18-65 of the students enrolled in the Guidance and Research Centers in Gebze and Darıca Districts in Kocaeli constitute the universe of the research. Using the G Power 3.1.9.4 program, the sample size calculated with a confidence interval of 0.05 and a power of 90% and a large effect size was calculated to be 16 for each group and a total of 32 caregiver studies. It is planned to reach 40 caregivers from each group and 80 caregivers in total, considering the parametric test assumptions and 10% sample loss. Randomization: After filling the pre-test questionnaires with the caregivers who agreed to participate in the research, it will be done by using the SPSS (24.0) statistical package program in the computer environment, taking into account the care burden, quality of life and psychological well-being scale scores. Inclusion Criteria; -Being between the ages of 18- 65, -Caring for a person with special needs for 6 months or more, -Having no physical dysfunction that would prevent doing yoga (COPD, septum deviation, etc.) -Having never done yoga before, -Refused to participate in the study -Speaking Turkish, -The caregiver has internet access, -The caregiver has a computer/tablet with a camera Exclusion criteria; - Having cognitive and musculoskeletal system, neuromuscular and chronic systemic diseases that prevent doing yoga, - Having had a surgical operation in the last 1 month, - Not being willing to participate in the study. Socio-demographic data and web-based yoga initiative were defined as independent variables. Scale total scores and sub-dimension total scores were defined as dependent variables. Socio-demographic Data Collection Form, Caregiver Burden Scale, Multidimensional Quality of Life Scale and Warwick-Edinburgh Mental Well-Being Scale will be applied to caregivers in the intervention and control groups included in the study. Informed consent will be obtained from caregivers participating in the study.

The yoga initiative to be applied to the intervention group; Yoga, which is mind-breath-body work; It includes meditation, pranayama (breath work), and asanas (yoga poses). The yoga practice will be applied by the researcher who has a RYT-200 Yoga Alliance yoga instructor certificate over the Zoom application in order to minimize the risk of infection, considering the COVID-19 pandemic period.

The content of the yoga practice consists of the following poses:

-Tadasana (Mountain pose), -Urdhvahastasana, -Uttanasana, -Ardha Uttanasana, -Plank, -Ashtang Pranam, -Bhujangasana (Mini cobra), -Adho Mukha Svanasana (Downward facing dog), -Vrksasana (Tree Pose), - Utthita Trikonasana (Triangle Pose), -Virabhadrasana I (Warrior I), -Virabhadrasana II (Warrior II), -Virabhadrasana I with Anjali Mudra (Hands Reverse Namaste), -Utkatasana (Chair Pose), -Salabhasana, -Paschimottanasana , -Dandasana, -Salamba Sarvangasana (Shoulder pose), -Ardha Urdhva Dhanurasana (Half Wheel Pose), -Reverse Warrior, -Child's pose, -Ananda Balasana (Happy baby), -Wipers, -Corpse Pose Evaluation of Data: While evaluating the data of the research, descriptive statistics (mean, std. deviation, median, etc.) for numerical variables and frequency distributions for categorical variables will be given. In the study, Kolmogorov Smirnov or Shapiro-Wilk normal distribution test will be used to examine the conformity of the variables to the normal distribution. Demographic data, total scores obtained from the scales in the experimental and control groups will be compared with the chi-square and t test. The difference between the experimental and control groups will be evaluated with an independent two-group t-test. The significance level will be accepted as 0.05. The power and effect size of the study will be calculated by regression analysis

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18- 65,
* Caring for an individual with special needs,
* Absence of cognitive and physical dysfunction that would prevent doing yoga,
* Agreeing to participate in the study and obtaining consent,
* Having never done yoga before
* Speaking Turkish,
* The caregiver has internet access,
* The caregiver has a computer/tablet/phone with a camera

Exclusion Criteria:

* Having cognitive and musculoskeletal system, neuromuscular and chronic systemic diseases that prevent doing yoga,
* Having had a surgical operation in the last 1 month,
* Not being willing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Caregiver Burden Scale | at 6 months
  The scoring of the 22-item scale is 1 (never), 2 (rarely), 3 (sometimes) and 4 (often) for each item. The total score of the scale ranges from 22 to 88. A maximum of 88 points can be obtained from the scale. The higher the score on the scale, the higher the burden of care is evaluated in the scale.
Multidimensional Quality of Life Scale (MILQ) | at 6 months
  The MILQ questionnaire is a 35-item scale addressing 9 sub-dimensions. The answers in the scale are numbered from 1 to 7. 1 is expressed as "not at all satisfied" and "7" is expressed as "very satisfied". The total score of the scale varies between 35-245. Higher scores represent better functional status.
Warwick-Edinburgh Mental Well-Being Scale | at 6 months
  It consists of 14 items, the scale is in 5-point Likert type and a minimum of 14 and a maximum of 70 points can be obtained from the scale. High scores from the scale indicate high mental (psychological) well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba ÖZDEMİR, PhD, Principal Investigator — Maltepe University; Gülendam KARADAĞ, PhD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Maltepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No